CLINICAL TRIAL: NCT04567654
Title: Assessment of the Topographic Relationship Between Mandibular Third Molars' Roots and the Covering Lingual Cortex in a Sample of Egyptian Population Using CBCT: An Observational Cross-Sectional Study
Brief Title: Assessment of the Relationship Between Mandibular Third Molars' Roots & the Covering Lingual Cortex Among Egyptian Population Using CBCT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Professor Hossam Kandil, Principal Investigator, Cairo University
Other Study IDs: RAD 7-1-1
Record Dates: First submitted 2020-09-17; First posted 2020-09-28 (Actual); Last update posted 2021-08-10 (Actual); Status verified 2020-09

CONDITIONS: Morphologic Change; Number of Roots
Keywords: mandibular third molars; mandibular third molars' roots; Lingual cortex; lingual cortex morphology; number of roots

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A cross-sectional study to assess the Topographic Relationship between Mandibular Third Molars' Roots and the Covering Lingual Cortex in a Sample of Egyptian Population using CBCT through retrospective data analysis

DETAILED DESCRIPTION:
Setting and Location:

The CBCT data of this study will be obtained from the CBCT database available at the Department of Oral and Maxillofacial Radiology, Faculty of Dentistry, Cairo University, Cairo, Egypt. Being a retrospective study, CBCT scans of Egyptian patients who have already been subjected to CBCT examination as part of their dental diagnosis and/or treatment planning will be included according to the proposed eligibility criteria.

Participants:

Based on sample size calculation, a sample of 304 mandibular third molar teeth belonging to Egyptian individuals will be examined. The selection of the scans to be included will be based on the following eligibility criteria

Eligibility criteria and selection method:

Inclusion criteria:

CBCT scans should show Mandibular third molars (Erupted &/or impacted) of Egyptian patients aging from 18 to 65 years old.

Mandibular third molars showing complete root formation.

Intact lingual cortex as well as intact mandibular third molars' roots.

CBCT scans of different fields of view (quadrant, single, or inter-arch) could be included as they show the mandibular third molars.

CBCT scans of a maximum of 0.4 mm voxel resolution will be included.

Exclusion criteria:

Mandibular third molars with developmental anomalies, external or internal root resorption, root canal calcification, previous root canal treatment, post restorations, and/or root caries.

Mandibular third molars with any pathology associated with and/or surrounding their roots.

CBCT images of sub-optimal quality or artifacts/high scatter interfering with proper assessment.

- Matching criteria and allocation ratio: Not applicable in the study.

Variables:

* Details about variable:

  1. Relationship between mandibular third molars' roots and covering lingual cortex
  2. Morphology of lingual cortex around mandibular third molars.
  3. Variation in number of roots of mandibular third molars.
* Data Sources / Measurements:

Retrospective Data Analysis will be performed after the CBCT images are pooled from the computer database.

Exposure parameters of the scans will vary depending on the individual patient's sizes

CBCT scans showing mandibular third molars with a maximum of 0.4 mm voxel size will be reviewed.

CBCT images will be analyzed using Planmeca Romexis® Viewer software, where the sagittal and coronal cross-sectional images will be oriented to be aligned with the long axis of the roots, together with the help of axial cross-sectional images for proper evaluation.

On the cross-sectional image, the relationship between mandibular third molars' roots and covering lingual cortex will be assessed at two levels (root apex and most lingual portion on apical one half) according to Emes classification: type A (non-contact), type B (contact), & type C (perforation).

The lingual cortex morphology around mandibular third molars' roots will also be assessed on the cross-sectional image according to the modified classification by Chan & Momin: Type U, undercut on the lingual side; Type P, parallel to the buccal plate; Type S, slanted with buccolingual width reduced on the lingual side, and Type R, round shape on the lingual side).

CBCT images will be interpreted by two oral radiologists independently; blinded from demographic data of the patients and from the results of each other.

Each radiologist will evaluate the images for assessment of number of roots, their relationship with covering the lingual cortex, and lingual cortex morphology. Then one of them will re-evaluate the images twice with two weeks interval between the two reading sessions.

Intra-observer and inter-observer and variability between the observers will be evaluated.

- Addressing potential sources of bias:

No source of bias. CBCT images will be interpreted by two oral and maxillofacial radiologists independently blinded from demographic data of the patients and from the results of each other.

Study Size:

The aim of this study is to detect the topographic relationship between mandibular third molars' roots and covering lingual cortex, lingual cortex morphology and variation in number of roots.

This power analysis used the relation between the lingual plate of bone and third molars' roots. Based upon Wang's results, the percentage of subjects with contact and perforation of lingual cortical plate was 72.8% using Alpha (α) level of (5%), acceptable margin of error = 5%, the minimum estimated sample size was 304 mandibular third molar teeth

Sample size calculation was performed using EPI Info 7.2.2.2.

Quantitative variables

- Handling of quantitative variables in analyses

Topographic relationship with the covering lingual cortex will be detected and categorically classified according to Emes classification: Type A (non-contact), Type B (contact), and type C (perforation).

The lingual cortex morphology will be detected and categorically classified according to modified Chan & Momin classification: (Type U, undercut on the lingual side; Type P, parallel to the buccal plate; Type S, slanted with bucco-lingual width reduced on the lingual side, and Type R, round shape on the lingual side).

The number of mandibular third molar roots will be numerically counted to estimate the variations in the Egyptian population.

Statistical methods:

- Statistical methods. Data will be statistically analyzed using IBM SPSS advanced statistics (Statistical Package for Social Sciences), version 23.0, Armonk, NY: IBM Corp. Numerical data will be described as mean and standard deviation or median and range. Categorical data will be described as numbers and percentages.

A p-value less than or equal to 0.05 will be considered statistically significant. All tests will be two-tailed.

ELIGIBILITY:
Inclusion Criteria:

* CBCT scans should show Mandibular third molars (Erupted &/or impacted) of Egyptian patients aging from 18 to 65 years old.
* Mandibular third molars showing complete root formation.
* Intact lingual cortex as well as intact mandibular third molars' roots.
* CBCT scans of different fields of view (quadrant, single, or inter-arch) could be included as they show the mandibular third molars.
* CBCT scans of a maximum of 0.4 mm voxel resolution will be included.

Exclusion Criteria:

* Mandibular third molars with developmental anomalies, external or internal root resorption, root canal calcification, previous root canal treatment, post restorations, and/or root caries.
* Mandibular third molars with any pathology associated with and/or surrounding their roots.
* CBCT images of sub-optimal quality or artifacts/high scatter interfering with proper assessment.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Egyptian population aging from 18 to 65 years old showing Mandibular third molars (Erupted &/or impacted) who have already been subjected to CBCT examination as part of their dental diagnosis and/or treatment planning
Sampling Method: Probability Sample
Enrollment: 304 (Estimated)
Dates: Start 2022-01-01 (Estimated); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-10-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of Topographic relationship Between mandibular third molars roots and the covering lingual cortex | 2 months
  The topographic relationship between roots and lingual cortex will undergo categorical assessment according to Emes classification: Type A (non-contact), Type B (contact), and type C (perforation)

SECONDARY OUTCOMES:
Assessment of lingual cortex morphology around roots of mandibular third molars | 2 months
  The lingual cortex morphology will undergo Categorical assessment according to modified Chan & Momin classification: (Type U, undercut on the lingual side; Type P, parallel to the buccal plate; Type S, slanted with bucco-lingual width reduced on the lingual side, and Type R, round shape on the lingual side).

OTHER OUTCOMES:
Assessment of variation in number of roots | 2 months
  The number of roots will be Numerically assessed

IPD SHARING:
Plan to Share IPD: Undecided
Still to decide whether to share it or not